CLINICAL TRIAL: NCT01215123
Title: Avastin in First Line Metastatic or Recurrent Breast Cancer. Retrospective Phase IV Study
Brief Title: An Observational Study of Avastin (Bevacizumab) in Patients With Metastatic Breast Cancer
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML25100
Record Dates: First submitted 2010-09-27; First posted 2010-10-06 (Estimated); Results first posted 2016-02-22 (Estimated); Last update posted 2016-02-22 (Estimated); Status verified 2016-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Bevacizumab: Participants received bevacizumab according to routine clinical practice until disease progression, unacceptable toxicity or withdrawal, along with taxane-based chemotherapy or in combination with other chemotherapy as prescribed.
  Interventions: Drug: Bevacizumab

INTERVENTIONS:
Drug: Bevacizumab — Participants received bevacizumab according to routine clinical practice until disease progression, unacceptable toxicity or withdrawal, along with taxane-based chemotherapy or in combination with other chemotherapy as prescribed.

SUMMARY:
This observational study will assess the median time of treatment duration and the safety of Avastin (bevacizumab) as first line treatment in patients with metastatic breast cancer. Data will be collected for approximately 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients with metastatic breast cancer in first line treatment who have completed treatment with Avastin

Exclusion Criteria:

* Patients not willing or unable to signed written consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients with first line treatment with Avastin
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2010-01; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (6):
- Argentina (6):
  - Buenos Aires
  - Capital Federal
  - La Pampa
  - Mar del Plata
  - Rosario
  - San Miguel de Tucumán

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study duration is January 2010 (first data collected) to July 2012 (last data collected). In this study, medical records of participants evaluated between 2008 and 2012 were reviewed.
Groups:
- Bevacizumab: Participants received bevacizumab according to routine clinical practice until disease progression, unacceptable toxicity or withdrawal, along with taxane-based chemotherapy or in combination with other chemotherapy as prescribed. Treatment continued for a maximum of 22 cycles.
Period: Overall Study
Arm/Group | Bevacizumab
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants
Arm/Group | Bevacizumab
Number analyzed (Participants) | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Disease Progression (TDP)
Description: Time to disease progression was defined as the time interval between first-line treatment onset and investigator-assessed disease progression. Disease progression was assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria and defined as at least a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: Up to a maximum of 36.4 months
Population: All enrolled participants
Measure: Median (Full Range); unit: months
Arm/Group | Bevacizumab
Number analyzed (Participants) | 28
months | 15.3 [2.6 to 36.4]

2. Secondary Outcome: Treatment Duration: Number of Bevacizumab Cycles
Description: Bevacizumab treatment duration in routine clinical practice was measured by the number of bevacizumab treatment cycles.
Time Frame: Up to a maximum of 36.4 months
Population: All enrolled participants
Measure: Median (Full Range); unit: cycles
Arm/Group | Bevacizumab
Number analyzed (Participants) | 28
cycles | 6 [1 to 22]

ADVERSE EVENTS:
Time Frame: Baseline up to 36.4 months
Description: All enrolled participants
Arm/Group | Bevacizumab
Serious Adverse Events (participants affected / at risk) | 10/28
Other Adverse Events (participants affected / at risk) | 23/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=28)
Asthenia (General disorders) | 5
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Bevacizumab (N=28)
Asthenia (General disorders) | 11
Edemas (General disorders) | 3
Cardiac event (not specified) (Cardiac disorders) | 2
Nausea (Gastrointestinal disorders) | 5
Vomits (Gastrointestinal disorders) | 2
Mucositis (Gastrointestinal disorders) | 4
Diarrhea (Gastrointestinal disorders) | 4
Liver event (not specified) (Hepatobiliary disorders) | 2
Neutropenia (Investigations) | 2
Anemia (Investigations) | 10
Myalgias (Musculoskeletal and connective tissue disorders) | 2
Arthralgias (Musculoskeletal and connective tissue disorders) | 3
Neuropathy (Nervous system disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 6
Hand-foot syndrome (Skin and subcutaneous tissue disorders) | 2
Allergy (Immune system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.